CLINICAL TRIAL: NCT01393769
Title: An Open, Single-centre Non-randomized Phase II Clinical Trial on Intra-arterial Chemotherapy With Melphalan for the Treatment of Retinoblastoma (RTB) in Advanced Intraocular Stage
Brief Title: Intra-arterial Chemotherapy With Melphalan for the Treatment of Retinoblastoma (RTB) in Advanced Intraocular Stage
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Only 5 subjects could be enrolled. Sample of 25 pat. not be achieved (rare disease).
Sponsor: Hospital Sant Joan de Deu (Other)
Collaborators: Fundació Sant Joan de Déu (Other); Hospital Universitari General de Catalunya (Other); Ministry of Health, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSJD-RTB-QTIA; 2009-010737-47 (EudraCT Number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-13 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma; RTB; Ocular tumour; Melfalan; Enucleation; Tumor of the eye; Eye; Ocular cancer; Ocular chemotherapy; Ophthalmic artery; Intra-arterial chemotherapy
MeSH Terms: conditions — Retinoblastoma; Eye Neoplasms | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melphalan (Experimental): Intra-arterial chemotherapy with melphalan, via direct administration by catheterization of the ophthalmic artery. Dosage range from 3 to 5 mg, depending of patient's weight and estimated tumour volume: a)3 mg for patients under 10 kg and tumour volume size under 1,5 cm3; b)5 mg for patients over 10 kg and tumour volume over 1,5 cm3; c)4 mg in all other situations(tumour volume over 1,5 cm3 in patients under 10 kg or tumour volume under 1,5 cm3 in patients over 10 kg).
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — The usual number of chemotherapy cycles will be 3. First treatment with Melphalan will be initiated as soon as possible, once the patients are selected for the study. Once the first treatment has been completed, day 0, successive treatments will be considered, second and third (days 21 and 42). In those cases in which some patients could be considered for an additional treatments after the third cycle, these will be administrated in intervals at least of 21 days.Dosage range from 3 to 5 mg, depending of patient's weight and estimated tumour volume.
  Other Names: Melfalan; Melfalan GlaxoSmithKline Inyectable

SUMMARY:
For selected cases with advanced Retinoblastoma (RTB) intraocular involvement(stage V of the Reese-Ellsworth classification) in which enucleation would usually be the standard therapeutic approach, in this project the investigators propose an alternative conservative treatment using intra-arterial chemotherapy with melphalan, via direct administration by catheterization of the ophthalmic artery.

DETAILED DESCRIPTION:
Retinoblastoma (RTB) is the most frequent tumour of the eye in early childhood and the commonest cancer in the first year of life. Approximately 60% of cases are sporadic and unilateral. Unilateral tumours are usually diagnosed in the advanced intraocular stage and the most frequent treatment prescribed is enucleation. This prevents disease progression but has an important visual risk, and also constitutes a mutilation, with potentially devastating psychological effects on patients and their relatives.

At diagnosis, patients affected with RTB and their relatives are faced with the important effects of this disease, such as a threat to life, although rare in developed countries, and the risk of losing their sight, which depends on the uni- or bilateral nature of the tumour, the topography of the tumour or tumours, and the still prevalent need for enucleation as a treatment. In fact, almost all advanced stage unilateral RTBs are treated with enucleation. In addition to the risk to life and the patient's sight associated with this treatment, it is also important to take into account the risk to the eye itself. For selected cases with advanced intraocular involvement (stage V of the Reese-Ellsworth classification) in which enucleation would usually be the standard therapeutic approach, in this project we propose an alternative conservative treatment using intra-arterial chemotherapy with melphalan, via direct administration by catheterization of the ophthalmic artery.

The treatment aims to preserve the eye ball and visual acuity as much as possible in these patients, and has been demonstrated to be extremely effective at achieving volumetric reduction of tumours, which permits, if necessary, the subsequent conservative treatment, mainly with brachytherapy for anterior tumours or thermotherapy with laser diode for posterior tumours. In cases of retinal detachment, significant volume reduction, such as that achieved after injection with melphalan would, in most cases, permit retinal reapplication that would favour visual prognosis.

This technique was first described by David H. Abramson in the Sloan-Kettering Cancer Center Memorial Hospital of New York (A Phase I/II Study of direct Intra-arterial (Ophthalmic Artery) Chemotherapy with Melphalan for Intraocular Retinoblastoma). Here, in this study we propose using this technique for the first time outside New York city, in our own clinical setting (Retinoblastoma Unit, affiliated to the Oncology Development Department and the Ophthalmology Department of the Sant Joan de Déu Hospital in Barcelona).

The attainment of positive results, in addition to those previously obtained by the New York project, could consolidate this treatment as an alternative to enucleation in most cases of advanced intraocular RTB, and open the way for the future indication of this technique in other stages of RTB.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral RTB.
2. Patients with advanced intraocular involvement, corresponding to Stage D of the International Classification , selected by the Tumour Committee of the Retinoblastoma Unit.

   By contrast to most other cancers, histological confirmation is contraindicated in RTB prior to onset of treatment and, in our study, any biopsy of the tumour practiced was considered as an exclusion criterion.
3. The only alternative to treatment is enucleation.
4. Over six months old at diagnosis and younger than six years old.
5. Informed consent of the parents or legal representative.

Exclusion Criteria:

1. Under 6 months old at diagnosis.
2. Impaired kidney function, with creatinine clearance lower than 80 mL/min/1.73m2 or serum creatinine higher than 0.7 mg/dL.
3. Impaired liver function, normal function being defined as presenting total bilirubin levels lower than 1.5 times the limit of normal for that age and ALT lower than 5 times the limit of normal for that age.
4. Patients with some type of coagulation disorder that could contraindicate the procedure or with a previous diagnosis of any thrombotic condition.
5. Congenital cerebral anomalies diagnosed previously or detected by angioresonance prior to treatment for extraocular involvement by RTB shown by image techniques, cerebrospinal fluid (CSF) cytology or cytomorphology of bone marrow aspirates (BMA), or positive expression of GD2 synthase in CSF or BMA.
6. Patients with heart disease, arterial hypertension, or diseases of the nervous system not referred to in point 5, or with active infections that the Anaesthesiology Service responsible for the procedure have studied and consider to contraindicate the procedure.
7. Not having been selected for intra-arterial chemotherapy through the ophthalmic artery for any other reason than those given by the Tumour Committee of the RTB Unit of the HSJD.
8. Concurrent administration of any other anti-cancer treatment.
9. Any surgical or non-surgical procedure that could have changed the structure of the eye and, therefore, facilitate risk of dissemination, including histological confirmation prior to treatment.
10. Participation in another clinical trial.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To assess the saving of eyes affected with RTB for patients who would have been candidates for enucleation. | From V1 (Baseline) to V14 (1+ year after last treatment)
  The primary endpoint will be the objective response to treatment determined by funduscopy and RetCam explorations, recorded as a percentage of partial response (PR) or complete response (CR) to the treatment administered.
The response will be evaluated as a function of tumoral volumetric size. | From V1 (Baseline) to V14 (+1 year after last treatment)
  The response will be evaluated as a function of tumoral volumetric size by comparing images obtained in successive funduscopy and RetCam explorations.

SECONDARY OUTCOMES:
To preserve visual acuity, by studying the affected eye after the third cycle of treatment. | V1 (Basal), V13 (day +52 to +60), V14 (+1 year after last treatment)
  The secondary endpoint studied will correspond to changes in visual acuity of the affected eye after the third cycle of treatment, assessed by a visual acuity study.
To modify the result of electroretinographic studies and visual evoked potentials after the third cycle of treatment. | V1 (Basal), V13 (day +52 to +60), V14 (+1 year after last treatment dosage)
  The secondary endpoint studied will correspond to changes in electroretinographic studies and visual evoked potentials after the third cycle of treatment
To evaluate the safety of the technique and medicinal product used, by studying the ophthalmologic and systemic adverse events. | Adverse events:on ongoing basis-assessed in each protocol visit / Laboratory test: V1 (Basal), V3&4 (day +1 to+10), V7&8 (day +22 to +31), V11&12 (day +43 to +52)
  The secondary safety endpoints studied will correspond to analytical changes in the CBC (essentially in the number of absolute neutrophils) and biochemistry analysis after 10 days of each treatment, and potential ophthalmologic side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Andreu Parareda, MD, Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Abramson DH, Dunkel IJ, Brodie SE, Kim JW, Gobin YP. A phase I/II study of direct intraarterial (ophthalmic artery) chemotherapy with melphalan for intraocular retinoblastoma initial results. Ophthalmology. 2008 Aug;115(8):1398-404, 1404.e1. doi: 10.1016/j.ophtha.2007.12.014. Epub 2008 Mar 14. PMID 18342944
- [Background] Aerts I, Pacquement H, Doz F, Mosseri V, Desjardins L, Sastre X, Michon J, Rodriguez J, Schlienger P, Zucker JM, Quintana E. Outcome of second malignancies after retinoblastoma: a retrospective analysis of 25 patients treated at the Institut Curie. Eur J Cancer. 2004 Jul;40(10):1522-9. doi: 10.1016/j.ejca.2004.03.023. PMID 15196536
- [Background] Apushkin MA, Apushkin MA, Shapiro MJ, Mafee MF. Retinoblastoma and simulating lesions: role of imaging. Neuroimaging Clin N Am. 2005 Feb;15(1):49-67. doi: 10.1016/j.nic.2005.02.003. PMID 15927860
- [Background] Brisse HJ, Lumbroso L, Freneaux PC, Validire P, Doz FP, Quintana EJ, Berges O, Desjardins LC, Neuenschwander SG. Sonographic, CT, and MR imaging findings in diffuse infiltrative retinoblastoma: report of two cases with histologic comparison. AJNR Am J Neuroradiol. 2001 Mar;22(3):499-504. PMID 11237973
- [Background] Chantada G, Doz F, Antoneli CB, Grundy R, Clare Stannard FF, Dunkel IJ, Grabowski E, Leal-Leal C, Rodriguez-Galindo C, Schvartzman E, Popovic MB, Kremens B, Meadows AT, Zucker JM. A proposal for an international retinoblastoma staging system. Pediatr Blood Cancer. 2006 Nov;47(6):801-5. doi: 10.1002/pbc.20606. PMID 16358310
- [Background] Chantada G, Fandino A, Manzitti J, Urrutia L, Schvartzman E. Late diagnosis of retinoblastoma in a developing country. Arch Dis Child. 1999 Feb;80(2):171-4. doi: 10.1136/adc.80.2.171. PMID 10325735
- [Background] Chantada GL, Dunkel IJ, de Davila MT, Abramson DH. Retinoblastoma patients with high risk ocular pathological features: who needs adjuvant therapy? Br J Ophthalmol. 2004 Aug;88(8):1069-73. doi: 10.1136/bjo.2003.037044. PMID 15258027
- [Background] Chantada GL, Fandino A, Mato G, Casak S. Phase II window of idarubicin in children with extraocular retinoblastoma. J Clin Oncol. 1999 Jun;17(6):1847-50. doi: 10.1200/JCO.1999.17.6.1847. PMID 10561224
- [Background] Chantada GL, Rossi J, Casco F, Fandino A, Scopinaro M, de Davila MT, Abramson DH. An aggressive bone marrow evaluation including immunocytology with GD2 for advanced retinoblastoma. J Pediatr Hematol Oncol. 2006 Jun;28(6):369-73. doi: 10.1097/00043426-200606000-00009. PMID 16794505
- [Background] Dunkel IJ, Aledo A, Kernan NA, Kushner B, Bayer L, Gollamudi SV, Finlay JL, Abramson DH. Successful treatment of metastatic retinoblastoma. Cancer. 2000 Nov 15;89(10):2117-21. doi: 10.1002/1097-0142(20001115)89:103.0.co;2-9. PMID 11066053
- [Background] Dunkel IJ, Gerald WL, Rosenfield NS, Strong EW, Abramson DH, Ghavimi F. Outcome of patients with a history of bilateral retinoblastoma treated for a second malignancy: the Memorial Sloan-Kettering experience. Med Pediatr Oncol. 1998 Jan;30(1):59-62. doi: 10.1002/(sici)1096-911x(199801)30:13.0.co;2-3. PMID 9371391
- [Background] Kaneko A, Suzuki S. Eye-preservation treatment of retinoblastoma with vitreous seeding. Jpn J Clin Oncol. 2003 Dec;33(12):601-7. PMID 14769836
- [Background] Kiribuchi M. [Retrograde infusion of anti-cancer drugs to ophthalmic artery for intraocular malignant tumors]. Nippon Ganka Gakkai Zasshi. 1966 Nov;70(11):1829-33. No abstract available. Japanese. PMID 6009660
- [Background] Moll AC, Imhof SM, Bouter LM, Kuik DJ, Den Otter W, Bezemer PD, Koten JW, Tan KE. Second primary tumors in patients with hereditary retinoblastoma: a register-based follow-up study, 1945-1994. Int J Cancer. 1996 Aug 7;67(4):515-9. doi: 10.1002/(SICI)1097-0215(19960807)67:43.0.CO;2-V. PMID 8759610
- [Background] Linn Murphree A. Intraocular retinoblastoma: the case for a new group classification. Ophthalmol Clin North Am. 2005 Mar;18(1):41-53, viii. doi: 10.1016/j.ohc.2004.11.003. PMID 15763190
- [Background] REESE AB, ELLSWORTH RM. The evaluation and current concept of retinoblastoma therapy. Trans Am Acad Ophthalmol Otolaryngol. 1963 Mar-Apr;67:164-72. No abstract available. PMID 13973597
- [Background] Rodriguez-Galindo C, Wilson MW, Haik BG, Merchant TE, Billups CA, Shah N, Cain A, Langston J, Lipson M, Kun LE, Pratt CB. Treatment of intraocular retinoblastoma with vincristine and carboplatin. J Clin Oncol. 2003 May 15;21(10):2019-25. doi: 10.1200/JCO.2003.09.103. PMID 12743157
- [Background] Shields CL, Shields JA, Baez K, Cater JR, De Potter P. Optic nerve invasion of retinoblastoma. Metastatic potential and clinical risk factors. Cancer. 1994 Feb 1;73(3):692-8. doi: 10.1002/1097-0142(19940201)73:33.0.co;2-8. PMID 8299091
- [Background] Shields CL, Shields JA, Minelli S, De Potter P, Hernandez C, Cater J, Brady L. Regression of retinoblastoma after plaque radiotherapy. Am J Ophthalmol. 1993 Feb 15;115(2):181-7. doi: 10.1016/s0002-9394(14)73922-4. PMID 8430727
- [Background] Shields JA, Parsons H, Shields CL, Giblin ME. The role of cryotherapy in the management of retinoblastoma. Am J Ophthalmol. 1989 Sep 15;108(3):260-4. doi: 10.1016/0002-9394(89)90116-5. PMID 2774035
- [Background] Muen WJ, Kingston JE, Robertson F, Brew S, Sagoo MS, Reddy MA. Efficacy and complications of super-selective intra-ophthalmic artery melphalan for the treatment of refractory retinoblastoma. Ophthalmology. 2012 Mar;119(3):611-6. doi: 10.1016/j.ophtha.2011.08.045. Epub 2011 Dec 22. PMID 22197434